CLINICAL TRIAL: NCT07009093
Title: Utility of a Mobile Application for Young Women With Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00119070; ONC-BRST-2401 (Other: Atrium Health)
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Cancer Distress
Keywords: Cancer-related Distress; Breast Cancer; Young Adult Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to the Mighty Pro Application (Experimental): Participants will be given access to the Mighty Pro Application for 12 months.
  Interventions: Other: Mighty Pro Application
- No Access to the Mighty Pro Application (No Intervention): Participants will not be given access to the Mighty Pro Application.

INTERVENTIONS:
Other: Mighty Pro Application — Access to Mighty Pro Application
  Arms: Access to the Mighty Pro Application

SUMMARY:
This study aims to evaluate the use of mobile technology as a communication tool among patients with breast cancer and measured its effect on patient-reported cancer-related distress, specifically focusing on young women as they often face unique challenges.

DETAILED DESCRIPTION:
This is a prospective, randomized, two stage study. The target population is adult females ≥ 18 and ≤ 45 years of age with breast cancer with a National Comprehensive Cancer Network (NCCN) Distress Thermometer score of distress score ≥ 4. The study will be conducted at Atrium Health Wake Forest Baptist Comprehensive Cancer Center (AHWFBCCC). The hypothesis is that the social connectivity via the Mighty Pro Application, as well as the educational components available in the application, will decrease patients' cancer-related distress. This study aims to evaluate the feasibility of implementing the Mighty Pro Application and measure its efficacy at reducing distress among young women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign an IRB-approved informed consent
* Age ≥ 18 and ≤ 45 years at the time of consent
* Female
* Established patient at Atrium Health Wake Forest Baptist Comprehensive Cancer Center (AHWFBCCC)
* Histological confirmation of any type and stage (0-IV) of breast cancer
* Screening (baseline) NCCN Distress Thermometer score ≥ 4
* Access to a mobile device for trial purposes and an active email address
* Ability to read and understand the English language. NOTE: The Mighty Pro Application is available in English only.
* As determined by the enrolling Investigator, ability of the participant to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

- None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Feasibility of Implementation of Mighty Pro App | 26 Weeks
  Binary variable indicating if at least one encounter with the application occurred for at least 80% of the weeks during the observation period. At the Participant level, the scale is either 0 (less than 80% utilization of the Mighty Pro App at least once per week during the 26-week observation period) or 1 (80% or greater utilization of the Mighty Pro App App at least once per week during the the 26-week observation period).
Stage 2: Efficacy of the Mighty Pro App | 26 Weeks
  Binary variable indicating if at least a 2-point improvement was achieved from baseline to 26 weeks. At the Participant level, the scale is either 0 (the study participant did not achieve at least a 2-point improvement from baseline to 26 weeks on the distress scale) or 1 (the study participant did achieve at least a 2-point improvement from baseline to 26 weeks on the distress scale). The distress scale ranges from 0 (no distress) to 10 (extreme distress).

SECONDARY OUTCOMES:
Efficacy of the Mighty Pro App in Improving Distress Scores | 52 Weeks
  Binary variable indicating if at least a 2-point improvement was achieved from baseline to 52 weeks. At the Participant level, the scale is either 0 (the study participant did not achieve at least a 2-point improvement from baseline to 52 weeks on the distress scale) or 1 (the study participant did achieve at least a 2-point improvement from baseline to 52 weeks on the distress scale). The distress scale ranges from 0 (no distress) to 10 (extreme distress).
Efficacy of the Mighty Pro App in Improving Distress Scores - Quantitative | 52 Weeks
  Quantitative distress scores collected for each participant and for each time point. For each Participant and each time point a quantitative measure will be collected ranging from 0 (no distress) to 10 (extreme distress).

CONTACTS AND LOCATIONS:
Overall Officials: Lejla Hadzikadic-Gusic, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Levine Cancer, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No